CLINICAL TRIAL: NCT01725867
Title: Comparing the Effect of Physical Therapy With Oral Appliance on Temporomandibular Disorder Related Myofascial Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Principal Investigator, National Taiwan University Hospital, National Taiwan University Hospital, National Taiwan University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201003038R
Record Dates: First submitted 2010-05-30; First posted 2012-11-14 (Estimated); Last update posted 2012-11-14 (Estimated); Status verified 2012-11

CONDITIONS: Temporomandibular Disorder
Keywords: temporomandibular joint disorder; myofascial pain; manual myofascial release; physical therapy; oral appliance
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PT program (Experimental): manual myofascial release for craniomandibular system for 30~40 minutes chin-in exercise within 10 minutes and as home exercise self-care education twice per week for 8 weeks
  Interventions: Other: PT program
- Splint group (Active Comparator): custom-made oral appliance: wear every night for 8 weeks, occasional drop is allowed self-care education
  Interventions: Device: oral appliance

INTERVENTIONS:
Other: PT program — manual myofascial release for craniomandibular system for 30~40 minutes chin-in exercise within 10 minutes and as home exercise self-care education twice per week for 8 weeks
  Arms: PT program
Device: oral appliance — custom-made oral appliance: wear every night for 8 weeks, occasional drop is allowed self-care education
  Arms: Splint group

SUMMARY:
the purpose of this study is to compare the effect of physical therapy (PT) program and oral appliance on patients with temporomandibular disorder (TMD)-related myofascial pain (MFP).

DETAILED DESCRIPTION:
The details of each intervention are listed as following:

* physical therapy program group (PT): manual myofascial release over craniomandibular system, chin-in exercise and self-care education
* oral appliance group (splint): custom-made stabilization splint and self-care education

ELIGIBILITY:
Inclusion Criteria:

* (1) 20-65 years old female, (2) diagnosed as MFP subtype of TMD according to Research Diagnostic Criteria for TMD (RDC/TMD), (3) pain duration over 3 month, (4) palpable taut band in masseter, (5) Asymmetrical pain intensity, (6) subsided symptoms of joint inflammation.

Exclusion Criteria:

* (1) traumatic TMD from external impact force, (2) history of traumatic cervical injury, (3) presence of systemic disease, (4) fibromyalgia, (5) co-interventions for cervical problems or TMD during study period, (6) signs of psychosomatic illness, (7) unwilling to be randomized, (8) unable to wear the splint or received intraoral myofascial release, (9)pregnancy.

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2010-06; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Pain status | 20 mins
  Visual analog scale (VAS) during functional activity and pressure pain threshold (PPT) of masseter taut bands

SECONDARY OUTCOMES:
range of motion (ROM) | 5 mins
  active and passive maximal mouth opening range
muscle strength | 5 mins
  maximal bite force
muscle endurance | 10 mins
  endurance of jaw closers
muscle stiffness | 10 mins
  stiffness of masseter taut band
Quality of life (QoL) | 15 mins
  quality of life measured by Short form-36 (SF-36) Taiwanese version

OTHER OUTCOMES:
stress | 5 mins
  Chinese 14-item perceived stress scale (PSS-14)

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan